CLINICAL TRIAL: NCT02864563
Title: Pan-genome Analysis of Neuroblastoma by Comparative Genomic Hybridization and Correlation With Pathology for the Diagnostic and the Prognostic Classification
Acronym: PHRCNB07
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IC 2007-09
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prospective cohort (Experimental): Experimental arm, prospective cohort
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — * Blood sample at diagnosis to evaluate MYCN amplification in plasma.
  * In case of NB with a MYCN amplification, blood samples are also collected during treatment and follow-up.

SUMMARY:
Neuroblastoma (NB) is characterized by its wide heterogeneity in clinical presentation and evolution. Recent retrospective studies have revealed by CGH-array that the overall genomic pattern is an important prognostic marker which might be taken into account for treatment stratification.

This protocol deals with a prospective analysis of the genomic profile established by CGH-array on the tumor samples obtained at the diagnosis of all the patients with NB in France, to obtain genomic profiles and being able to determine their prognostic impact in the various protocols of treatment. The objective of this study will be a better therapeutic stratification in the future trials, studies or protocols of treatment.

DETAILED DESCRIPTION:
After diagnosis of Neuroblastoma (NB) or Ganglioneuroblastoma :

* Frozen tumor sample (cell content ≥60%) must be sent for genomic profile determination by CGH-array,
* Blood sample at diagnosis must be sent to evaluate MYCN amplification in plasma,
* In case of NB with a MYCN amplification, blood sample during treatment and follow-up must be sent.

ELIGIBILITY:
Inclusion Criteria:

1. Neuroblastoma or Ganglioneuroblastoma defined by INSS criteria (Brodeur et al. 1993)
2. Age < 18 years
3. Availability of tumoral sample obtained at diagnosis, prior chemotherapy with tumor cell content ≥ 60%
4. Inclusion in 4 months following the diagnosis
5. All patients treated in French centers (SFCE) for Neuroblastic tumour, including those participate in national or international protocols.

7. Written informed consent 8. Patients with French Social Security in compliance with the French law relating to biomedical research.

Exclusion Criteria:

1. Chemotherapy or radiotherapy before taking tumour samples
2. Refusal of the parents or the legal representatives

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 560 (Actual)
Dates: Start 2008-10-04 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2023-07 (Actual)

PRIMARY OUTCOMES:
Progression-Free survival | 3 years
  Time between patient diagnosis and tumoral progression or relapse or death. Correlation with the genomic profile established by CGH-array.

SECONDARY OUTCOMES:
Progression at metastatic location-Free survival | 3 years
  Time between patient diagnosis and progression/ relapse at metastatic location or death.
  Correlation with the genomic profile established by CGH-array.
Overall-Free survival | 3 years
  Time between patient diagnosis and death.Correlation with the genomic profile established by CGH-array.

CONTACTS AND LOCATIONS:
Overall Officials: Gudrun Shleiermacher, MD, PhD, Principal Investigator — Institut Curie
Locations (27):
- France (27):
  - Hôpital Nord Amiens, Amiens
  - Chu Angers, Angers
  - Chr R.Pellegrin, Bordeaux
  - CHU MORVAN Brest, Brest
  - CHR CAEN, Caen
  - Chu Bocage, Dijon
  - Chu Grenoble, Grenoble
  - Chu Lille, Lille
  - Hopital de La Mere Et de L'Enfant Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Hopital D'Enfants de La Timone, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHR MONCOUSU Nantes, Nantes
  - CHU Nice Hôpital L'Archet 2, Nice
  - Institut Curie, Paris
  - Hôpital Armand TROUSSEAU, Paris
  - Hôpital Jean Bernard de la Milétrie, Poitiers
  - Höpital Americain Reims, Reims
  - CHR Hôpital Sud Rennes, Rennes
  - Hôpital Charles Nicolle ROUEN, Rouen
  - Chr Felix Guyon, Saint-Denis
  - CHU SAINT-ETIENNE Hôpital Nord, Saint-Priest-en-Jarez
  - Hôpital Hautepierre Strasbourg, Strasbourg
  - Hôpital des Enfants Toulouse, Toulouse
  - CHU TOURS Hôpital Clocheville, Tours
  - Hopital Des Enfants Nancy, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets with interested researchers, educators or clinicians. Materials generated under the project will be disseminated in accordance with Institut Curie policies.
Time Frame: Data requests can be submitted starting 9 months after article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).